CLINICAL TRIAL: NCT06692803
Title: Real-World Treatment Patterns and Outcomes Among Patients With Chronic Myeloid Leukemia in Earlier Lines of Therapy (ABL-2022-03)
Brief Title: Real-World Treatment Patterns and Outcomes Among Patients With Chronic Myeloid Leukemia in Earlier Lines of Therapy
Acronym: ABL-2022-03
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A0US04
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- First Treatment Cohort: Patients newly diagnosed with CML who received first treatment with imatinib, dasatinib, nilotinib, or bosutinib.
- Second Treatment Cohort: Patients from first treatment cohort with a subsequent line of therapy (i.e., second treatment) with imatinib, dasatinib, nilotinib, bosutinib, or ponatinib.

SUMMARY:
This was a retrospective, non-interventional, observational cohort study using Optum's de-identified Clinformatics® Data Mart Database. Adult patients newly diagnosed with chronic myeloid leukemia (CML) treated with tyrosine kinase inhibitors (TKIs) were identified using the Optum database and classified into the following cohorts:

* First treatment cohort: Patients newly diagnosed with CML who received first treatment with a TKI.
* Second treatment cohort: Patients from first treatment cohort with a subsequent line of therapy (i.e., second treatment) with a TKI.

The observation period spanned from the start of data availability (i.e., 01 January 2007) to the earliest of end of data (i.e., 30 June 2022), end of continuous health plan enrollment, or death (if available). The index date was defined as the first treatment initiation for the first treatment TKI cohort and as the second treatment initiation for the second treatment TKI cohort. The baseline period consisted of the 6 months prior to the index date. The follow-up period started on the index date and ended at the earliest of end of observation period or hematopoietic stem cell transplantation (HSCT).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who initiated their first treatment with imatinib, dasatinib, nilotinib, or bosutinib (conditional on Food and Drug Administration (FDA) approval dates) with 6 months continuous health plan enrollment prior to the first prescription fill date.
* Patients with 2 or more diagnoses for CML (adult as of the first diagnosis for CML).
* Patients had index date on or after first CML diagnosis.
* Patients had no diagnoses for CML remission/relapse prior to index date.
* Patients had no gastrointestinal stomach tumor (GIST) or chronic myelomonocytic leukemia (CMML) at any time.
* Patients had no medical claims associated with a clinical trial during the baseline period.
* Patients had no hematopoietic stem cell transplantation (HSCT) during the baseline period.
* Patients had no CML-related chemotherapy treatments for accelerated phase (AP)/blast crisis (BC) during the baseline period.
* First treatment cohort:

  * Patients started first treatment for CML with imatinib, dasatinib, nilotinib, or bosutinib in 2012 or later.
  * Patients had no HSCT during the first treatment baseline period.
  * Patients had no CML-related chemotherapy treatment for AP/BC during the first treatment baseline period.
* Second treatment cohort:

  * Patients started second treatment for CML with imatinib, dasatinib, nilotinib, or bosutinib in 2012 or later.
  * Patients had no HSCT from the first treatment baseline period up to second treatment initiation.
  * Patients had no CML-related chemotherapy treatment for AP/BC from the first treatment baseline period up to second treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 2043 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Treatment Patterns | Up to approximately 10 years
  Tyrosine kinase inhibitor (TKI) treatment management patterns in CML patients on first line or second line TKI were assessed.

SECONDARY OUTCOMES:
Proportion of Days Covered (PDC) | Up to approximately 10 years
  PDC was defined as the number of days of medication covered divided by the number of calendar days during the study period. The study period spanned from index date to the next line of therapy initiation (switch), hematopoietic stem cell transplantation (HSCT), initiation of a CML-related chemotherapy for accelerated phase (AP)/blast crisis (BC) (day prior to HSCT/CML chemotherapy) or last supply day if treatment gap ≥ 90 days, whichever occurred first. The index date was defined as the first treatment initiation for the first treatment cohort and as the second treatment initiation for the second treatment cohort.
Number of Patients per PDC Category | Up to approximately 10 years
  PDC was defined as the number of days of medication covered divided by the number of calendar days during the study period. The study period spanned from index date to the next line of therapy initiation (switch), HSCT, initiation of a CML-related chemotherapy for AP/BC (day prior to HSCT/CML chemotherapy) or last supply day if treatment gap ≥ 90 days, whichever occurred first. The index date was defined as the first treatment initiation for the first treatment cohort and as the second treatment initiation for the second treatment cohort.
  PDC categories included:
  * PDC (%) ≤ 50%
  * PDC (%) ≤ 70%
  * PDC (%) ≥ 80%
  * PDC (%) > 90%
Time to Treatment Discontinuation | Up to approximately 10 years
Time to Treatment Switch | Up to approximately 10 years
Time to First Treatment Interruption | Up to approximately 10 years
Time to First Dose Reduction | Up to approximately 10 years
Rate of Treatment Discontinuation | Months 1, 3, 6, 9, 12, 18, and years 2, 3, 4
Rate of Treatment Switching | Months 1, 3, 6, 9, 12, 18, and years 2, 3, 4
Rate of Treatment Interruption | Months 1, 3, 6, 9, 12, 18, and years 2, 3, 4
Rate of Dose Reduction | Months 1, 3, 6, 9, 12, 18, and years 2, 3, 4
Number of Patients With Non-optimal Treatment (NOPT) | Up to approximately 10 years
  Three categories of NOPT were defined:
  1. Base Case: NOPT was defined as 1) treatment switch ≤ 6 months post-index, 2) temporary treatment interruption/dose reduction ≤6 months post-index followed by treatment switch ≤12 months post-index, or 3) PDC ≤50%.
  2. Sensitivity 1: NOPT was defined as 1) treatment switch ≤ 6 months post-index, 2) temporary treatment interruption/dose reduction ≤6 months post-index followed by treatment switch ≤12 months post-index, or 3) PDC ≤70%.
  3. Sensitivity 2: NOPT was defined as treatment switch ≤ 6 months post-index.
  Index date was defined as the first treatment initiation for the first treatment cohort and as the second treatment initiation for the second treatment cohort.
Number of Patients With NOPT by First Generation TKI | Up to approximately 10 years
  Three categories of NOPT were defined:
  1. Base Case: NOPT was defined as 1) treatment switch ≤ 6 months post-index, 2) temporary treatment interruption/dose reduction ≤6 months post-index followed by treatment switch ≤12 months post-index, or 3) PDC ≤50%.
  2. Sensitivity 1: NOPT was defined as 1) treatment switch ≤ 6 months post-index, 2) temporary treatment interruption/dose reduction ≤6 months post-index followed by treatment switch ≤12 months post-index, or 3) PDC ≤70%.
  3. Sensitivity 2: NOPT was defined as treatment switch ≤ 6 months post-index.
  Index date was defined as the first treatment initiation for the first treatment cohort and as the second treatment initiation for the second treatment cohort.
Number of Patients With NOPT by Second Generation TKI | Up to approximately 10 years
  Three categories of NOPT were defined:
  1. Base Case: NOPT was defined as 1) treatment switch ≤ 6 months post-index, 2) temporary treatment interruption/dose reduction ≤6 months post-index followed by treatment switch ≤12 months post-index, or 3) PDC ≤50%.
  2. Sensitivity 1: NOPT was defined as 1) treatment switch ≤ 6 months post-index, 2) temporary treatment interruption/dose reduction ≤6 months post-index followed by treatment switch ≤12 months post-index, or 3) PDC ≤70%.
  3. Sensitivity 2: NOPT was defined as treatment switch ≤ 6 months post-index.
  Index date was defined as the first treatment initiation for the first treatment cohort and as the second treatment initiation for the second treatment cohort.
All-cause Healthcare Resource Utilization (HRU) per Patient per Year in NOPT Patients Compared to Reference Subgroup | 2 years
  The reference subgroup was defined based on the following treatment adherence and persistence criteria denoting potential indicators of TKI treatment success based on observations from the clinical practice: (1) high treatment adherence (defined as PDC >90%) with no observed treatment discontinuation anytime post-index; or (2) high treatment adherence (defined as PDC >90%) with treatment discontinuation occurring >12 months post-index.
  All-cause HRU included:
  * Inpatient admission
  * Inpatient days
  * Emergency department visits
  * Outpatient visits
CML-related HRU per Patient per Year in NOPT Patients Compared to Reference Subgroup | 2 years
  The reference subgroup was defined based on the following treatment adherence and persistence criteria denoting potential indicators of TKI treatment success based on observations from the clinical practice: (1) high treatment adherence (defined as PDC >90%) with no observed treatment discontinuation anytime post-index; or (2) high treatment adherence (defined as PDC >90%) with treatment discontinuation occurring >12 months post-index.
  All-cause HRU included:
  * Inpatient admission
  * Inpatient days
  * Emergency department visits
  * Outpatient visits
All-cause Direct Healthcare Costs per Patient per Year in NOPT Patients Compared to Reference Subgroup | 2 years
  The reference subgroup was defined based on the following treatment adherence and persistence criteria denoting potential indicators of TKI treatment success based on observations from the clinical practice: (1) high treatment adherence (defined as PDC >90%) with no observed treatment discontinuation anytime post-index; or (2) high treatment adherence (defined as PDC >90%) with treatment discontinuation occurring >12 months post-index.
  All-cause direct healthcare costs included:
  * Total medical costs
  * Inpatient costs
  * Outpatient costs
  * Emergency department costs
CML-related Direct Healthcare Costs per Patient per Year in NOPT Patients Compared to Reference Subgroup | 2 years
  The reference subgroup was defined based on the following treatment adherence and persistence criteria denoting potential indicators of TKI treatment success based on observations from the clinical practice: (1) high treatment adherence (defined as PDC >90%) with no observed treatment discontinuation anytime post-index; or (2) high treatment adherence (defined as PDC >90%) with treatment discontinuation occurring >12 months post-index.
  All-cause direct healthcare costs included:
  * Total medical costs
  * Inpatient costs
  * Outpatient costs
  * Emergency department costs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States